CLINICAL TRIAL: NCT00375050
Title: Neuroprotective Treatment of Refractory Schizophrenia With Riluzole 01T-432
Brief Title: Treatment of Refractory Schizophrenia With Riluzole
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13175
Record Dates: First submitted 2006-09-08; First posted 2006-09-12 (Estimated); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Schizophrenia; Schizoaffective
MeSH Terms: conditions — Schizophrenia | interventions — Riluzole

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Riluzole (Experimental)
  Interventions: Drug: Riluzole
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Riluzole
  Other Names: Rilutek
  Arms: Riluzole
Drug: Placebo — placebo
  Arms: Placebo

SUMMARY:
The proposed study would evaluate the benefits of riluzole add-on treatment to patients with schizophrenia who are already receiving medications, but still experience symptoms. Neuroprotective medication riluzole is currently approved for treatment of amyotrophic lateral sclerosis (Lou Gehrig's disease), a severe neurological illness. Due to its unique mechanism of action, riluzole, if effective in helping the symptoms of schizophrenia, would open novel directions in treatment of schizophrenia.

DETAILED DESCRIPTION:
Schizophrenia is perhaps one of the most debilitating illnesses. Over the past years there has been limited improvement in the efficacy of the medications used to treat this disorder. In particular, the currently available antipsychotic drugs have small efficacy against negative symptoms and cognitive impairment associated with schizophrenia. This is critical considering that both negative symptoms and cognitive deficits contribute significantly to social and vocational impairment in schizophrenic patients. Furthermore, current treatment can not always provide satisfactory control of positive symptoms. While various extracellular neurotransmitter systems (dopamine, 5HT, GABA, etc. ) have been explored as targets for antipsychotic treatment, a substantial body of evidence suggests that neurodegenerative intracellular processes might be responsible for some of the symptoms of schizophrenia, resulting in cytopathic effects or inadequate cellular functioning. Some of these processes may be triggered by excitotoxic influence of neurotransmitters (i.e. glutamate). As many neuroleptic agents currently in use have some neuroprotective properties it is possible to speculate that medications with primarily neuroprotective mode of action might be of additional help in treatment of schizophrenia.

Huntington's disease patients who in its advanced form exhibit some symptoms similar to that of psychotic illness, have, in a recent small (n=9) open label study with a neuroprotective drug riluzole, shown a temporary improvement in not only motor function, but also cognitive, and behavioral functioning (Seppi 2001).

Based on all of the above, it seems possible to expect improvement in symptoms of schizophrenia with neuroprotective agents such as riluzole.

Riluzole is the only effective medication approved for use in ALS (amyotrophic lateral sclerosis, Lou Gehrig's disease) which is one of the most severe and rapidly progressing neurodegenerative illnesses that affects motor neurons in the brain and spinal cord. A subset of ALS is inherited and involves more than 70 different mutations in the antioxidant enzyme superoxide dismutase (SOD) thereby contributing to reduced antioxidative defense against oxidative injury. This results in increased reactive oxygen species level in several organs/tissues while the bulk of symptomatology is related to degeneration in the subset of CNS neurons. Although riluzole is effective in both humans and the transgenic mouse model of familial ALS where it slows decrease in motor power, its exact neuroprotective mechanism of action is not known. Various studies suggest that riluzole might exert some of its beneficial effect by inhibition of glutamate release, inhibition of voltage-gated Na+ channels, but also intracellularly by inhibiting of protein kinase C (PKC), enzyme that was linked to oxidative neuronal injury. Although riluzole is generally well tolerated, side effects can occur and are mostly related to gastrointestinal problems, hepatotoxicity and asthenia.

This 14 week study would evaluate the benefits of riluzole add-on treatment to patients with schizophrenia on neuroleptics with refractory symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Men or women with a diagnosis of schizophrenia or schizoaffective disorder as defined by DSM- IV criteria.
* Age between 18 and 65. Special attention will be placed on selective enrolling of patients 18-25 to assess that they have been exposed to adequate medication trials (minimum two medications) for sufficient length of time.
* During the 3 months prior to study entry, the patient must not have been an inpatient in a hospital for longer than 4 weeks (cumulative hospitalizations) due to worsening of psychiatric illness (although could have been participating in an inpatient research protocol).
* Patients able to comprehend and satisfactorily comply with the protocol requirements;
* Patients with a PANSS total score of 60 or higher and a score of 4 (moderate) or higher on two or more of the following PANSS items: delusions, hallucinatory behavior, conceptual disorganization or suspiciousness.
* CGI scale rating of at least mildly ill, but not greater than severely ill.
* For women only: The patient must be non-pregnant, non-lactating, or has undergone tubal ligation, bilateral oophorectomy or hysterectomy; or the patient must be at least one year post menopausal; or the patient a) has negative urine or serum pregnancy test (Beta HCG) and b) agrees to reliably practice contraception throughout the study.

Exclusion Criteria:

* Primary psychiatric diagnosis other than schizophrenia or schizoaffective disorder.
* Patients who have had psychosurgery
* Recent (< 3 weeks) change in antipsychotic regimen
* Presence of clinically significant somatic disease that requires frequent changes in medications or that could be aggravated by taking riluzole (i.e. severe liver illness)
* Currently receiving treatment with potentially hepatotoxic drugs (e.g. allopurinol, methyldopa, sulfasalazine)
* HIV positive, as assessed by blood testing (in part to avoid subjects with possible brain HIV infection and to avoid rare complications of rarely occurring riluzole induced neutropenia)
* Patients who pose immediate or significant enough risk for suicide or harm for others as assessed by the study MD.
* Pregnant or nursing women, or women of childbearing potential who do not use adequate contraception or who are judged to be unreliable in their use of contraception (because there is not enough experience with riluzole use in nursing or pregnant women)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2002-05; Primary Completion 2006-08-29 (Actual); Study Completion 2006-08-29 (Actual)

PRIMARY OUTCOMES:
PANSS (Positive and Negative Syndrome Scale) | 12 weeks
SANS (Scale for the Assessment of Negative Symptoms) | 12 weeks
CGI- Clinical Global Impression Scale | 12 weeks
Calgary Depression Scale: To assess mood symptoms in psychotic patients | 12 weeks
Neuropsychological tests: | 12 weeks
Computerized Working Memory Task | 12 weeks
Verbal Fluency | 12 weeks
HVLT-Hopkins Verbal Learning Test | 12 weeks
DSST-Digit Symbol Substitution Test | 12 weeks
Continuous performance test | 12 weeks
CANTAB- Cambridge Neuropsychological Test Automated Battery | 12 weeks
AIMS (abnormal involuntary movement scale), EPS (extrapyramidal symptom) assessment, Barnes akathisia scale, Simpson Angus scale | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Zoran Zimolo, MD, Ph.D., Principal Investigator — Yale University
Locations (1):
- Yale Department of Psychiatry, New Haven, Connecticut, United States